CLINICAL TRIAL: NCT02305095
Title: Genomic Analysis of the Enhanced Response to Heart Failure Therapy in African Americans
Brief Title: Genomic Response Analysis of Heart Failure Therapy in African Americans
Acronym: GRAHF-2
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Dennis M. McNamara, MD, MS, Professor of Medicine and Director, Center for Heart Failure Research, University of Pittsburgh
Other Study IDs: 3648634; MD009118-01 (Other Grant/Funding Number: National Institute on Minority Health and Health Disparities)
Record Dates: First submitted 2014-09-25; First posted 2014-12-02 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — isosorbide-hydralazine combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and DNA banked at baseline.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- GNB3 TT: All subjects with the GNB3 TT genotype for the polymorphism at position 825 (T/C). They will be initiated on therapy with FDC I/H, followed for 2 years and response to therapy quantified by a composite score (CS).
  Interventions: Drug: FDC I/H
- GNB3 C: All subjects with at least one copy of the GNB3 C allele which includes both subjects homozygous for the 825C allele (GNB3 CC genotype) and subjects who are heterozygous (GNB3 TC genotype).They will be initiated on therapy with FDC I/H, followed for 2 years and response to therapy quantified by a composite score (CS).
  Interventions: Drug: FDC I/H

INTERVENTIONS:
Drug: FDC I/H — All subjects in both groups will be initiated on drug, FDC I/H with dose titrated up to target doses based on clinical guidelines
  Other Names: BiDil

SUMMARY:
The response to therapy with a fixed dose combination of isosorbide dinitrate and hydralazine (FDC I/H) is enhanced in African Americans with heart failure and reduced ejection fraction (HFrEF) when compared to similar white cohorts. This study will seek to confirm the previous genetic sub-study from AHeFT which suggested a functional polymorphism of guanine nucleotide binding protein beta polypeptide 3 subunit (GNB3), C825T in exon 10, influences the therapeutic efficacy of FDC I/H. This study will initiate treatment with FDC I/H in 500 self designated African American subjects with systolic heart failure. They will be followed for up to two years on therapy. Clinical outcomes (survival, heart failure hospitalizations, and change in quality of life) on FDC I/H will be compared by GNB3 genotype subset. The hypothesis to be confirmed is that subjects homozygous for the T allele (those with the GNB3 TT genotype which is present in approximately 50% of black subjects) demonstrate enhanced therapeutic benefit from FDC I/H.

DETAILED DESCRIPTION:
The response to therapy with a fixed dose combination of isosorbide dinitrate and hydralazine (FDC I/H) is enhanced in African Americans with heart failure and reduced ejection fraction (HFrEF) when compared to similar white cohorts. Despite the clear survival benefits of treatment with FDC I/H in the African American Heart Failure Trial (AHeFT), the drug is prescribed in only 25% of black subjects who would potentially benefit.

In terms of the enhanced response evident in the A-HeFT investigation, race is likely a marker of differences in genomic background. Genetic variation of the G protein beta sub unit GNB3 has been studied extensively for its role in hypertension. A polymorphism exists at position 825 (T/C) which is functionally silent but tightly linked to a splicing variant resulting in a truncated protein. The GNB3 T haplotype is far more prevalent in blacks and associated with low renin hypertension. Evaluation of 350 subjects in the genetic sub-study of AHeFT suggests that the GNB3 TT genotype, found in 50% of African Americans but only 10-15% of whites, was linked to an enhanced therapeutic response to FDC I/H. This investigation will evaluate the hypothesis that the GNB3 TT genotype is a marker of enhanced therapeutic response to FDC I/H in African Americans with HFrEF.

The study will enroll a cohort of 500 African Americans with HFrEF, initiate therapy with FDC I/H and follow them for up to two years. Subjects will be genotyped at entry for the GNB3 polymorphism and response to therapy compared by genotype. Therapeutic response will be quantified using the composite score, the primary endpoint of AHeFT, which incorporates mortality, heart failure hospitalizations, and a change in quality of life (QoL) score at six months.

Aim 2 will do a similar analysis of response to therapy by GNB3 genotype using improvement in left ventricular end diastolic diameter (LVEDD) or left ventricular ejection fraction (LVEF) by echocardiogram after six months on therapy as the outcomes measure. Aim 3 will use admixture analysis to determine first how global ancestry (the % African ancestral DNA for an individual) impacts on the outcome measures of drug response, and how the global ancestry acts as a modifier for the effect of GNB3.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older
2. History of heart failure with an LVEF (less than OR equal to) < 0.35 for at least 6 months OR an LVEF < 0.45 with left ventricular internal end diastole (defined by a diameter of more than 2.9 cm per square meter of body surface area OR more than 6.5 cm on the basis of echocardiography). ** Echo must be done within 6 months of enrollment**
3. New York Heart Association (NYHA) Class II-IV
4. Background heart failure therapy that includes angiotensin converting enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARBs), and beta blockers (BBs) for at least 3 months (or documentation of intolerance to ACEi/ARBs and BBs)
5. Self-designated race as African American or black (would include subjects whose country of origin was outside the USA such as Africa, the Caribbean, or Central America).

Exclusion Criteria:

1. History of intolerance to either nitrates or hydralazine
2. Treatment with the combination of hydralazine and nitrates for the previous 3 months
3. Revascularization or myocardial infarction within last 90 days
4. Received cardiac resynchronization therapy (CRT) AND did not have an assessment of cardiac function documenting an LVEF < 35% (less than OR equal to 35%) at least 90 days post CRT
5. Presence of clinically significant valvular heart disease, hypertrophic or restrictive cardiomyopathy, active myocarditis, or uncontrolled hypertension. (Note that uncontrolled hypertension is defined as blood pressure consistently greater than 160 mmHg systolic and 95 mmHg diastolic)
6. Women who are currently pregnant, planning on becoming pregnant in the next two years, or those who do not agree to prevent pregnancy.
7. Subjects who are on continuous home inotropes, a left ventricular assist device, or who are post cardiac transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with systolic heart failure who are self designation as African Americans are potentially eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Composite score (CS) no units. (survival, heart failure hospitalization, and change in the raw quality of life score on the Minnesota Living with Heart Failure Questionnaire) | 2 years
  The CS combines three outcome variables into a single "score". Composite score adds points for survival over 2 years of follow up (death at any time yields -3 points, survival to end of study results in 0), heart failure hospitalization over 2 years of follow up (yes at any time results in -1 point, no results in 0), and the change in the raw quality of life score on the Minnesota Living with Heart Failure Questionnaire from entry to 6 months (change of ten units or greater=increase +2, decrease-2; change 5 to 9= increase+1, decrease -1; change < 5 units for the raw score yields 0 points). The CS will range from -6 to +2 for each patient.

SECONDARY OUTCOMES:
Survival | 2 years
  Comparison of survival on therapy by GNB3 genotype
Survival free from heart failure hospitalization | 2 years
  Comparison of event free survival by GNB3 genotype.
Change in Quality of Life Assessment by Minnesota Living with Heart Failure Questionnaire | 6 months
  Evaluate the change in the raw score of the Quality of Life questionnaire by GNB3 genotype.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis McNamara, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (19):
- United States (19):
  - University of Alabama Medical Center, Tuscaloosa, Alabama
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois of Chicago, Chicago, Illinois
  - Tulane University Heart and Vascular Institute, New Orleans, Louisiana
  - Ochsner, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachsetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Rutgers University Health Center, Newark, New Jersey
  - Montefiore Medical Center Bronx New York, The Bronx, New York
  - MetroHealth System, Cleveland, Ohio
  - Temple University Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia